CLINICAL TRIAL: NCT00492531
Title: Treatment of Pulmonary Hypertension and Sickle Cell Disease With Sildenafil Therapy
Brief Title: Sildenafil Therapy for Pulmonary Hypertension and Sickle Cell Disease
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Subjects on drug were more likely to have severe pain crises requiring hospitalization.
Sponsor: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Principal Investigator, Mark Gladwin, Professor and Chair of Medicine, National Heart, Lung, and Blood Institute (NHLBI)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 070177; 07-H-0177 (Other: IRB Approval number , NHLBI)
Record Dates: First submitted 2007-06-26; First posted 2007-06-27 (Estimated); Results first posted 2011-06-06 (Estimated); Last update posted 2016-01-06 (Estimated); Status verified 2015-12

CONDITIONS: Sickle Cell Disease; Pulmonary Hypertension
Keywords: Interventional Study; 6-Minute Walk; Sickle Cell Anemia; Sildenafil/Viagra; Tricuspid Regurgitant Velocity; Sickle Cell Disease; Pulmonary Hypertension
MeSH Terms: conditions — Anemia, Sickle Cell; Hypertension, Pulmonary | interventions — Sildenafil Citrate; Phosphodiesterase 5 Inhibitors; Sugars

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Sildenafil (Experimental): There was a balancing of treatment group assignment across Tricuspid Regurgitant Jet velocity(TRV)measured on Echo.
  Interventions: Drug: Sildenafil
- Placebo (Placebo Comparator): There was a balancing of treatment group assignment across Tricuspid Regurgitant Jet velocity(TRV)measured on Echo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Sildenafil — Oral Sildenafil 20mg three times daily for 6 weeks,followed by 40mg three times daily for 4 weeks followed by 80mg three times daily for 6 weeks.
  Other Names: phosphodiesterase-5(PDE5) inhibitor
  Arms: Sildenafil
Drug: Placebo — Placebo 20mg three times daily for 6 weeks,followed by 40mg three times daily for 4 weeks followed by 80mg three times daily for 6 weeks.
  Other Names: Sugar pill
  Arms: Placebo

SUMMARY:
This study will examine whether the drug sildenafil can lower blood pressure in the pulmonary artery (the blood vessel that leads from the heart to the lungs) in patients with sickle cell disease and pulmonary hypertension (high blood pressure in the lungs). It will see if this treatment can reduce disease complications, such as shortness of breath, pain crisis, pneumonia, and increase survival.

Patients 12 years of age and older with sickle cell disease and pulmonary hypertension may be eligible for this study. Participants are randomly assigned to receive sildenafil or placebo (sugar pill) for 16 weeks. Before starting treatment, patients have baseline studies, including a pregnancy test for females of childbearing age; a chest x-ray; pulmonary function tests to measure how much air the patient can breathe in and out; an echocardiogram (heart ultrasound); a 6-minute walk test to measure exercise capacity; a quality-of-life assessment and a pain inventory. Patients with moderate to severe pulmonary hypertension undergo heart catheterization to evaluate the severity of hypertension before beginning sildenafil therapy.

During treatment, patients are monitored with the following:

* Blood tests: weeks 6, 10 and 16.
* Echocardiogram: weeks 6 and 16.
* 6-minute walk test: weeks 6, 10 and 16.
* Measurements of weight, blood pressure and heart rate: weeks 6, 10 and 16.
* Pregnancy test for women of childbearing age: weeks 6, 10 and 16.
* Pain questionnaire once a day for a week: weeks 6 and 1.0
* Quality-of-life questionnaire: week 16.
* Heart catheterization: week 16 for patients with moderate to severe hypertension.

At the end of the 16-week period, patients may opt to continue to receive sildenafil and monitoring in an open-label phase of the study for up to 1 year.

DETAILED DESCRIPTION:
Sickle cell disease (SCD) is an autosomal recessive disorder and the most common genetic disease affecting African-Americans. Approximately 0.15 percent of African-Americans are homozygous for sickle cell disease, and 8 percent have sickle cell trait. Acute pain crisis, acute chest syndrome (ACS), and pulmonary hypertension are common complications of sickle cell anemia. Pulmonary hypertension (PH) has now been identified as a marker of mortality in adults with sickle cell disease. Sildenafil has been proven beneficial in pulmonary hypertension (PH) and recent phase I/II studies from the intramural National Institutes of Health (NIH) suggest it is well tolerated and efficacious in the SCD population. Furthermore, a number of recent studies have suggested that nitric oxide (NO) based therapies may have a favorable impact on sickle red cells at the molecular level and could improve the abnormal microvascular perfusion that is characteristic of sickle cell anemia.

The project has 3 distinct components:

1. Screening Phase. Approximately 1000 subjects with sickle cell disease will be screened. Assessments will include historical and laboratory data, Doppler echocardiogram, 6-minute walk test, plasma/serum, and DNA for banking.
2. Main Interventional Trial. The randomized, double-blind, placebo controlled phase is designed to determine the effects of 16 weeks of Sildenafil therapy on exercise endurance, cardiopulmonary hemodynamic parameters and symptoms in this patient population. The open-label follow-up phase is designed to provide up to an additional year of Sildenafil therapy to subjects who completed the randomized, double-blind phase.
3. Observational Follow-up Study. Screened patients who do not qualify for participation in the main interventional trial may be contacted every 6-12 months for up to 3 years to assess major disease-related complications, including mortality.

ELIGIBILITY:
• Eligibility based on the following inclusion and exclusion criteria.

INCLUSION CRITERIA:

Screening Phase:

* Males or females, greater than or equal to 12 years of age and less than or equal to 70 years of age.
* Diagnosis of sickle cell disease (including, but not limited to SS, SC, SD, or S-beta zero thalassemia).
* Provision of informed consent and, where applicable, assent.

Observational Follow-up Study:

* Satisfaction of screening criteria.
* In the opinion of the investigator, ability to maintain follow-up contact.
* Failure to satisfy the eligibility requirements of the Main Interventional Trial (MIT) OR discontinuation/completion of the MIT/Open-label Follow-up Phase.
* Provision of informed consent and, where applicable, assent.

Main Interventional Trial:

* Males or females, 12 years of age or older and less than or equal to 70 years of age.
* Female subjects, on a reliable method of birth control or not physically able to bear children.
* Electrophoretic documentation of sickle cell disease (including, but not limited to SS, SC, SD, or S-beta zero thalassemia).
* At least mild pulmonary hypertension with TRV greater than or equal to 2.7 m/sec by echocardiogram.
* Six-minute walk distance of 150-500 m.
* In the opinion of the investigator, able to complete the protocol scheduled assessments during the 16-week, double-blind phase.
* Provision of informed consent and, where applicable, assent.
* Subjects with systemic hypertension must be on a stable antihypertensive regimen for greater than or equal to 90 days and a stable dose for greater than or equal to 30 days.

EXCLUSION CRITERIA:

Current pregnancy or lactation.

Any one of the following medical conditions:

* Stroke within the last six weeks.
* Diagnosis of pulmonary embolism within the last three months.
* History of retinal detachment or retinal hemorrhage in the last 6 months.
* Non-arteritic anterior ischemic optic neuropathy (NAION) in one or both eyes.
* History of sustained priapism requiring medical or surgical treatment, unless currently impotent or on transfusion program within the last two years.
* Any unstable (chronic or acute) condition that in the opinion of the investigator will prevent completion of the study.

Subjects taking nitrate-based vasodilators (including, but not limited to nicorandil [available in the UK only]), prostacyclin (inhaled, subcutaneous or intravenous) or endothelin antagonists. Subjects taking calcium channel blockers will be allowed to participate if they are on a stable dose for greater than or equal to 3 months.

Left ventricular ejection fraction (LVEF) less than 40 percent or clinically significant ischemic, valvular or constrictive heart disease: LVEF less than 40 percent or SF less than 22 percent.

Subjects in other research studies with investigational drugs (with the exception of hydroxyurea) unless the other trial has been approved by the walk-PHaSST Executive Committee for co-participation.

Acute or chronic impairment (other than dyspnea), limiting the ability to comply with study requirements (in particular with 6MWT), e.g., angina pectoris, intermittent claudication, symptomatic hip osteonecrosis.

Tonsillectomies for sleep apnea within 3 months prior to randomization. Active therapy for pulmonary hypertension, including prostacyclin analog, endothelin-1 antagonist, or PDE-5 inhibitor.

Protease inhibitor therapy for HIV treatment Subjects taking potent CYP3A4 inhibitor therapy (e.g., itraconazole, ritonavir, ketoconazole) Subjects who are anticoagulated and have proliferative retinopathy (unless they have had ophthalmologist recommended intervention (e.g., phototherapy) or have been cleared by the ophthalmologist to participate in the study.

Subjects with systolic blood pressure greater than or equal to 140 mmHg OR diastolic blood pressure greater than or equal to 90 mmHg.

Ages: 12 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 74 (Actual)
Dates: Start 2007-06; Primary Completion 2009-09 (Actual); Study Completion 2009-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mark T Gladwin, M.D, Principal Investigator — Professor of Medicine: Chief, Pulmonary, Allergy and Critical CRE Medicine: Director, Hemostasis and Vascular Biology Research Institute; University of Pittsburgh School of Medicine
Locations (9):
- United States (8):
  - Children's Hospital, Oakland, Oakland, California
  - University of Colorado, Denver, Colorado
  - Howard University Hospital, Washington D.C., District of Columbia
  - University of Illinois at Chicago, Chicago, Illinois
  - Johns Hopkins University, Baltimore, Maryland
  - National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland
  - Albert Einstein College of Medicine, The Bronx, New York
  - Childrens Hospital, Pittsburgh, Pittsburgh, Pennsylvania
- Imperial College London and Hammersmith Hospital, London, United Kingdom

REFERENCES:
- [Background] Castro O. Systemic fat embolism and pulmonary hypertension in sickle cell disease. Hematol Oncol Clin North Am. 1996 Dec;10(6):1289-303. doi: 10.1016/s0889-8588(05)70401-9. PMID 8956017
- [Background] Sutton LL, Castro O, Cross DJ, Spencer JE, Lewis JF. Pulmonary hypertension in sickle cell disease. Am J Cardiol. 1994 Sep 15;74(6):626-8. doi: 10.1016/0002-9149(94)90760-9. No abstract available. PMID 8074054
- [Background] Verresen D, De Backer W, Vermeire P. Pulmonary hypertension and sickle hemoglobinopathy. Chest. 1990 Oct;98(4):1042. doi: 10.1378/chest.98.4.1042a. No abstract available. PMID 2209119
- [Derived] D'Alessandro A, Nouraie SM, Zhang Y, Cendali F, Gamboni F, Reisz JA, Zhang X, Bartsch KW, Galbraith MD, Espinosa JM, Gordeuk VR, Gladwin MT. Metabolic signatures of cardiorenal dysfunction in plasma from sickle cell patients as a function of therapeutic transfusion and hydroxyurea treatment. Haematologica. 2023 Dec 1;108(12):3418-3432. doi: 10.3324/haematol.2023.283288. PMID 37439373
- [Derived] Liggett LA, Cato LD, Weinstock JS, Zhang Y, Nouraie SM, Gladwin MT, Garrett ME, Ashley-Koch A, Telen MJ, Custer B, Kelly S, Dinardo CL, Sabino EC, Loureiro P, Carneiro-Proietti AB, Maximo C; NHLBI Trans-Omics for Precision Medicine (TOPMed) Consortium; Reiner AP, Abecasis GR, Williams DA, Natarajan P, Bick AG, Sankaran VG. Clonal hematopoiesis in sickle cell disease. J Clin Invest. 2022 Feb 15;132(4):e156060. doi: 10.1172/JCI156060. PMID 34990411
- [Derived] Page GP, Kanias T, Guo YJ, Lanteri MC, Zhang X, Mast AE, Cable RG, Spencer BR, Kiss JE, Fang F, Endres-Dighe SM, Brambilla D, Nouraie M, Gordeuk VR, Kleinman S, Busch MP, Gladwin MT; National Heart, Lung, and Blood Institute (NHLBI) Recipient Epidemiology Donor Evaluation Study-III (REDS-III) program. Multiple-ancestry genome-wide association study identifies 27 loci associated with measures of hemolysis following blood storage. J Clin Invest. 2021 Jul 1;131(13):e146077. doi: 10.1172/JCI146077. PMID 34014839
- [Derived] Sinha AA, Adusumilli T, Cohen HW, Nouraie M, Little J, Manwani D. Splenectomy is not associated with a higher tricuspid regurgitant jet velocity in people with sickle cell anemia. Pediatr Blood Cancer. 2019 Oct;66(10):e27928. doi: 10.1002/pbc.27928. Epub 2019 Jul 19. PMID 31322833
- [Derived] Gladwin MT, Barst RJ, Gibbs JS, Hildesheim M, Sachdev V, Nouraie M, Hassell KL, Little JA, Schraufnagel DE, Krishnamurti L, Novelli E, Girgis RE, Morris CR, Berman Rosenzweig E, Badesch DB, Lanzkron S, Castro OL, Taylor JG 6th, Goldsmith JC, Kato GJ, Gordeuk VR, Machado RF; walk-PHaSST Investigators and Patients. Risk factors for death in 632 patients with sickle cell disease in the United States and United Kingdom. PLoS One. 2014 Jul 2;9(7):e99489. doi: 10.1371/journal.pone.0099489. eCollection 2014. PMID 24988120
- [Derived] Nouraie M, Lee JS, Zhang Y, Kanias T, Zhao X, Xiong Z, Oriss TB, Zeng Q, Kato GJ, Gibbs JS, Hildesheim ME, Sachdev V, Barst RJ, Machado RF, Hassell KL, Little JA, Schraufnagel DE, Krishnamurti L, Novelli E, Girgis RE, Morris CR, Rosenzweig EB, Badesch DB, Lanzkron S, Castro OL, Goldsmith JC, Gordeuk VR, Gladwin MT; Walk-PHASST Investigators and Patients. The relationship between the severity of hemolysis, clinical manifestations and risk of death in 415 patients with sickle cell anemia in the US and Europe. Haematologica. 2013 Mar;98(3):464-72. doi: 10.3324/haematol.2012.068965. Epub 2012 Sep 14. PMID 22983573
- [Derived] Sachdev V, Kato GJ, Gibbs JS, Barst RJ, Machado RF, Nouraie M, Hassell KL, Little JA, Schraufnagel DE, Krishnamurti L, Novelli EM, Girgis RE, Morris CR, Rosenzweig EB, Badesch DB, Lanzkron S, Castro OL, Taylor JG 6th, Hannoush H, Goldsmith JC, Gladwin MT, Gordeuk VR; Walk-PHASST Investigators. Echocardiographic markers of elevated pulmonary pressure and left ventricular diastolic dysfunction are associated with exercise intolerance in adults and adolescents with homozygous sickle cell anemia in the United States and United Kingdom. Circulation. 2011 Sep 27;124(13):1452-60. doi: 10.1161/CIRCULATIONAHA.111.032920. Epub 2011 Sep 6. PMID 21900080
- [Derived] Machado RF, Barst RJ, Yovetich NA, Hassell KL, Kato GJ, Gordeuk VR, Gibbs JS, Little JA, Schraufnagel DE, Krishnamurti L, Girgis RE, Morris CR, Rosenzweig EB, Badesch DB, Lanzkron S, Onyekwere O, Castro OL, Sachdev V, Waclawiw MA, Woolson R, Goldsmith JC, Gladwin MT; walk-PHaSST Investigators and Patients. Hospitalization for pain in patients with sickle cell disease treated with sildenafil for elevated TRV and low exercise capacity. Blood. 2011 Jul 28;118(4):855-64. doi: 10.1182/blood-2010-09-306167. Epub 2011 Apr 28. PMID 21527519
- See also: NIH Clinical Center Detailed Web Page — http://clinicalstudies.info.nih.gov/detail/B_2007-H-0177.html

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects with Sickle cell hemoglobinopathy were recruited from 10 centers(9 in United States and 1 in United Kingdom)
Groups:
- Sildenafil: Subjects received oral sildenafil 20 mg three times daily for six weeks, followed by 40 mg three times daily for four weeks, followed by 80 mg three times daily for six weeks (as tolerated).
- Placebo: Subjects received matching oral dose of placebo 20 mg three times daily for six weeks, followed by 40 mg three times daily for four weeks, followed by 80 mg three times daily for six weeks (as tolerated).
Period: Overall Study
Arm/Group | Sildenafil | Placebo
Started | 37 | 37
Completed | 15 (Of 15 subjects who completed study, 13 were enrolled in Open label.) | 14 (Of 14 subjects who completed study, 13 were enrolled in Open label.)
Not Completed | 22 | 23
Not completed — Withdrawn(More than one reason selected) | 22 | 23

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Sildenafil | Placebo | Total
Number analyzed (Participants) | 37 | 37 | 74
Age, Continuous [Mean (Standard Deviation); unit: years] | 47 (13) | 44 (14) | 45 (13)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 23 | 23 | 46
  Male | 14 | 14 | 28
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 32 | 37 | 69
  Unknown or Not Reported | 5 | 0 | 5
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 36 | 37 | 73
  White | 0 | 0 | 0
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 1 | 0 | 1
6 minute walk [Mean (Standard Deviation); unit: Meters] — The distance walked in six minute was used to assess the exercise capacity of the patient at baseline.
  Meters | 381 (75) | 386 (75) | 383 (75)
Tricuspid regurgitant jet velocity (TRV) [Mean (Standard Deviation); unit: m/s] — Tricuspid regurgitant jet velocity was measured by transthoracic Doppler Echocardiography.
  m/s | 3.0 (0.5) | 3.0 (0.3) | 3.0 (0.3)

OUTCOME MEASURES:

1. Secondary Outcome: Change From Baseline in Pulmonary Hypertension at Week 16 as Assessed by Tricuspid Regurgitant Jet Velocity
Description: Secondary outcome measure was change from baseline in Pulmonary hypertension at week 16 as assessed by Tricuspid regurgitant jet velocity(TRV). Tricuspid regurgitant jet velocity was measured by transthoracic Doppler Echocardiography.
Time Frame: 16 weeks
Measure: Mean (Standard Deviation); unit: meters/second
Arm/Group | Sildenafil | Placebo
Number analyzed (Participants) | 37 | 37
meters/second
  Baseline | 3.1 (0.5) | 3.0 (0.3)
  Week 6 | 3.2 (0.7) | 2.9 (0.3)
  Week 16 | 2.9 (0.5) | 2.9 (0.3)

2. Secondary Outcome: Borg Dyspnea Score
Description: Borg dyspnea score was used to measure the level of severity of breathlessness perceived by the patient before and after 6 minute walk. The severity is measured on a 10 point scale with 0= nothing at all and 10=maximum severity of breathlessness.
Time Frame: baseline to 16 weeks
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Sildenafil | Placebo
Number analyzed (Participants) | 37 | 37
Score on a scale
  Baseline | 2.5 (2.1) | 2.1 (2.0)
  Week 6 | 3.4 (2.3) | 1.8 (1.3)
  Week 10 | 2.7 (2.0) | 2.7 (1.7)
  Week 16 | 2.0 (1.6) | 2.8 (2.4)

3. Secondary Outcome: Brain Natriuretic Peptide(BNP)Levels.
Time Frame: 16 weeks
Measure: Mean (Standard Deviation); unit: pg/dl
Arm/Group | Sildenafil | Placebo
Number analyzed (Participants) | 35 | 35
pg/dl
  Baseline | 2.3 (0.6) | 2.0 (0.6)
  Week 6 | 2.4 (0.4) | 2.0 (0.7)
  Week 10 | 2.3 (0.5) | 2.2 (0.6)
  Week 16 | 2.5 (0.7) | 2.3 (0.6)

4. Primary Outcome: Change in Exercise Capacity as Assessed by 6 Minute Walk.
Description: The primary outcome measure was change in exercise capacity assessed by 6 minute walk distance in meters from baseline to 16 weeks. Subjects without a week 16 assessment had their last observation carried forward.
Time Frame: Baseline to week 16/Imputed last visit.
Population: All efficacy and safety analyses were conducted on the intent-to-treat (ITT) population, defined as all randomized subjects, regardless of therapy received. Pre-defined imputation rules:A value of 0 meters was imputed for subjects who died during the MIT.Subjects without a week 16 assessment had their last observation carried forward (LOCF).
Measure: Mean (Standard Deviation); unit: meters
Arm/Group | Sildenafil | Placebo
Number analyzed (Participants) | 37 | 37
meters | -16 (20) | -7 (20)
Statistical Analysis 1: Comparison: Sildenafil vs Placebo; Test type: Superiority or Other; p = 0.70, ANCOVA; 6 minute walk was based on ANCOVA model with treatment as a fixed effect and 6 minute walk distance, TRV stratum and study site as covariate; Mean Difference (Net) = -9, 95% CI 2-sided [-56 to 38]

ADVERSE EVENTS:
Time Frame: Safety assessments were conducted at baseline, weeks 6, 10 (excluding echocardiography), and 16.
Description: Treatment group differences in AEs and SAEs were evaluated via Cochran-Mantel-Haenszel chi-square tests, controlling for TRV stratum. The study was stopped early due to the higher percentage of subjects experiencing an SAE in the sildenafil arm as compared to the placebo arm.
Arm/Group | Sildenafil | Placebo
Serious Adverse Events (participants affected / at risk) | 17/37 | 8/37
Other Adverse Events (participants affected / at risk) | 30 | 28
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Sildenafil (N=37) | Placebo (N=37)
Acute chest syndrome (Blood and lymphatic system disorders) | 1 | 3
Anemia (Blood and lymphatic system disorders) | 2 | 1
Sickle cell anemia with crisis (Congenital, familial and genetic disorders) | 13 | 5
Bronchitis (Infections and infestations) | 1 | 0
Lower respiratory tract infection (Infections and infestations) | 1 | 0
Hyperkalemia (Metabolism and nutrition disorders) | 0 | 2
Hypertension (Vascular disorders) | 0 | 1
Hypotension (Vascular disorders) | 1 | 0
Atrial fibrillation (Cardiac disorders) | 1 | 0
Congestive Cardiac failure (Cardiac disorders) | 1 | 0
Vitreous hemorrhage (Eye disorders) | 1 | 0
Pyrexia (General disorders) | 1 | 0
Traumatic brain injury (Injury, poisoning and procedural complications) | 1 | 0
Suicide attempt (Psychiatric disorders) | 1 | 0
Acute pulmonary edema (Respiratory, thoracic and mediastinal disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected / at risk:
Term (organ system) | Sildenafil | Placebo
SCA with Crisis (Congenital, familial and genetic disorders) | 18/37 | 13/37
Headache (Nervous system disorders) | 13/37 | 4/37
Musculoskeletal and connective tissue disorders (Musculoskeletal and connective tissue disorders) | 5/37 | 6/37
Blood and Lymphatic system disorders (Blood and lymphatic system disorders) | 4/37 | 6/37
Eye disorders (Eye disorders) | 5/37 | 4/37
Blurred vision (Eye disorders) | 5/37 | 1/37
General Disorders and administration site conditions (General disorders) | 6/37 | 3/37
Infections and infestations (Infections and infestations) | 5/37 | 14/37

LIMITATIONS AND CAVEATS:
As a result of early termination due to safety findings, the study was underpowered to assess the effects of sildenafil therapy on the predetermined efficacy endpoints.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No